CLINICAL TRIAL: NCT04738968
Title: Cochlear Implant for Young Children and One Deaf Ear
Brief Title: Cochlear Implantation for Young Single-sided Deaf Children
Acronym: CICADE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Cochlear (Industry); Agentschap Innoveren & Ondernemen (VLAIO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S57318
Record Dates: First submitted 2014-12-08; First posted 2021-02-04 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Deafness Unilateral
Keywords: auditory rehabilitation; cochlear implant; single-sided deafness
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the test or the control group
Masking Description: It is known whether the child has a cochlear implant or not
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cochlear implant for single-sided deafness (Experimental): Children with single-sided deafness, cochlear implant in the deaf ear
  Interventions: Device: Cochlear implant
- Control single-sided deafness (No Intervention): Children with single-sided deafness, no intervention
- Control normal hearing (No Intervention): Children with normal hearing, no intervention

INTERVENTIONS:
Device: Cochlear implant — A cochlear implant is standard care for profoundly deaf persons. It enables hearing through electrical stimulation of the auditory nerve.
  Arms: Cochlear implant for single-sided deafness

SUMMARY:
Children with profound sensorineural unilateral hearing loss (UHL) lag behind in spoken language, cognition, spatial hearing, and academic performance compared to normal hearing (NH) children. Until recently children with UHL were not remediated, thereby assuming that the normal ear would provide sufficient sensory cues for speech understanding. However, this is not true. Because of the difference between the two ears they have difficulty localizing sounds and understanding speech in noise. Such auditory deprivation leads to more global changes in neurocognitive function. It is expected that a cochlear implant in the deaf ear will provide the necessary cues for hearing with two ears. The main objective of this research project is to fundamentally investigate language, cognitive, and spatial/binaural hearing longitudinally in children with unilateral deafness who receive a cochlear implant and age-matched peers.

DETAILED DESCRIPTION:
The main objective of the research project is to fundamentally investigate spatial and binaural hearing in a group of children with a normal hearing ear (NH) and a cochlear implant (CI) longitudinally in order to understand the relationship between sensory experience and auditory cortex plasticity. This relationship is most striking during infancy when changes in sensory input can have profound effects on the functional organization of the developing cortex. Recent studies in the auditory system have revealed the remarkably adaptive nature of sensory processing and provided important insights into the way in which cortical circuits are shaped by experience and learning. The binaural system processes and integrates differences in phase (low frequencies) or intensity (high frequencies) between sounds arriving at the left and right ear and this process goes on from birth up to adulthood. It is expected that cochlear implantation will promote normal or near-normal spatial-hearing skills in children with UHL and that intervention at 2 years of age yields the best conditions for (near-) normal development of cognition, spoken language, balance, and psychopathology, outcomes which will be monitored annually too.

Fifteen NH-CI children, aged 2 or younger, will receive a cochlear implant. This device has already been provided to over 400.000 bilaterally profoundly deaf persons worldwide and is considered a standard treatment. The novelty of the present studies lies in the treatment of unilaterally deaf children with a cochlear implant. Because of the cost of this device, the Belgian government does not reimburse a CI for children with unilateral hearing impairment, which is why a study is done to demonstrate its effectiveness. The 15 devices are provided by Cochlear. While the sample size may seem small, providing the device (25.000€ a piece) and some follow-up (mapping and/or remediation) are a large investment for Cochlear Ltd. The children will act as their own control (tested with and without CI) when possible. In addition, at the start of the research project the NH-CI children will be age-matched with 15 normal hearing children (NH-NH), and with 15 children with unilateral hearing loss without a CI (NH - x). Care will be taken to control for as many other factors as possible (e.g. other disabilities, parental and socioeconomic characteristics, ..).

It is hypothesized that the children with UHL and a CI (NH-CI) will outperform children without intervention (NH-x) because of access to bilateral input, and that provision at a very young age will result in near-normal binaural processing in the following years and hence better auditory/neuro/cognitive processing and learning in general. After cochlear implantation, the children will be followed up in terms of language development, cognitive development, binaural hearing, and academic achievements.

ELIGIBILITY:
Inclusion Criteria:

* profoundly hearing impaired in one ear
* normal hearing in contralateral ear

Exclusion Criteria:

none

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Spoken language comprehension | Every 6 months between 2nd and 5th birthday
  The Schlichting Test for Receptive Language is a language comprehension test for children aged 2 to 7 years. Results are reported as an age-referenced language comprehension quotient based on the total score.
Spoken language production (young children) | Every 6 months between 2nd and 5th birthday
  The Schlichting Test for Expressive Language is a language production test for children aged 2 to 7 years. Results are reported as age-referenced language quotients for each subtest, namely (1) expressive vocabulary, (2) morphosyntactic skills, (3) auditory memory, (4) pseudoword repetition, (5) story telling.
Spoken language production (older children) | Yearly from the age of 5, until study completion (average period: 2 years)
  The Clinical Evaluation of Language Fundamentals (CELF-4-NL) is a language test for children aged 5 to 18 years. Results are reported as age-referenced scores for some of the subtests, namely (1) word structure, (2) sentence repetition, (3) sentence production, (4) word categories, (5) phonologic awareness.
Spatial speech perception in noise | Yearly from the age of 4, until study completion (average period: 3 years)
  Speech perception in noise is measured for three spatial conditions using the LittleLINT speech material (numbers 1-10). Results are reported for each condition as the speech reception threshold, i.e. the level (in decibel signal-to-noise ratio, dB SNR) at which 50% of the speech is understood. Children with a CI are tested both with and without their device.
Sound localization | Yearly from the age of 4, until study completion (average period: 3 years)
  Sound localization is assessed in a 9-loudspeaker setup with 15° degrees spacing between the loudspeakers. The stimulus is a 1-second broadband telephone sound. Results are reported as the mean absolute error, i.e. the average difference (in degrees) between the active loudspeaker and the child's response. Children with a CI are tested both with and without their device.

SECONDARY OUTCOMES:
Cognitive development (young children) | Every 6 months until the age of 3.5 years
  The Bayley Scales of Infant and Toddler Development (Bayley-III-NL) is a developmental test for children aged 0 to 4 years and includes cognitive, language, and motor assessment scales. Results are reported as an age-referenced cognitive quotient for the cognitive scale.
Cognitive development (older children) | At 4 and 6 years of age (i.e. twice in total)
  The Wechsler Preschool & Primary Scale of Intelligence (WPPSI-III-NL) is a cognitive development test for children aged 2 to 8 years. Results are reported as age-referenced composite scores or intelligence quotients (IQs), namely (1) full IQ, (2) verbal IQ, (3) performance IQ, (4) processing speed.
Functional balance | Yearly from the age of 4, until study completion (average period: 3 years)
  The Balance scale of the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) provides a nine-item screening for balance problems, for children aged 4 to 22 years. Results are reported as an age-referenced standard score.
Speech perception with the cochlear implant alone | At clinical visits after the age of 3, on average 2 times per year, until study completion (average period: 4 years)
  In the group of single-sided deaf children with a cochlear implant, speech perception using only the implant is measured using the Lilliput speech materials. The sound is streamed directly to the implant to avoid contribution from the normal hearing ear. Results are reported as speech perception scores (in percentages).

OTHER OUTCOMES:
Binaural integration and cortical symmetry | One EEG session after the age of 5
  Using electroencephalography (EEG), the cortical reorganization effect of single-sided deafness is assessed in a subsample of children with compared to without cochlear implant. Cortical onset responses and bilateral auditory steady-state responses (ASSRs) are used to derive a measure for both cortical symmetry and binaural integration.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid van Wieringen, PhD, Principal Investigator — KU Leuven; Irem Adalilar, MSc, Study Director — KU Leuven
Locations (4):
- Belgium (4):
  - Antwerp University Hospital, Antwerp
  - GZA Hospitals, Antwerp
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven